CLINICAL TRIAL: NCT05822336
Title: The Relationship Between Pain Intensity and Intramuscular Injection
Brief Title: Duration of IM Injection and Pain Intensity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Leman Şenturan, Prof. Dr., Biruni University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: BiruniUn
Record Dates: First submitted 2023-03-17; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Pain Measurement
Keywords: Intramusculer Injection; Nurse; Pain Intensity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Repeated measure
Who Masked: Participant
Masking Description: Single blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): In this group, the duration of IM injections was 40 seconds. The drug was the same for both groups, Clindamycin 600 mg/4 ml intramuscularly.
  Interventions: Other: Duration of Intramuscular Injections
- Active arm (No Intervention): In this group, the duration of IM injections was 10 seconds. The drug was the same for both groups, Clindamycin 600 mg/4 ml intramuscularly.

INTERVENTIONS:
Other: Duration of Intramuscular Injections — This study was a single-group crossover clinical trial, where each participant acted as their own control. Two intramuscular injections into the right and left Dorsal Gluteal Region (DRG) were recorded for each participant. One was administered by a nurse, according to the unit's routine, and took 5 seconds to complete. A day after, the same nurse gave the other injection in the opposite DGR, taking 40 seconds to administer. The five-second injections were considered the control group, while the 40 seconds injections were the intervention group. The order of interventions was randomized. The pain level was determined and recorded immediately after each injection.
  Arms: Experimental arm

SUMMARY:
This study was a single-group crossover clinical trial, where each participant acted as their own control. The study aimed to describe the relationship between perceived pain and the duration of intramuscular injections

DETAILED DESCRIPTION:
The study was a single-group crossover clinical trial, where each participant acted as their own control. The study sample included 50 patients aged 25 to 55 who met the inclusion criteria of signing an informed consent form and requiring administration of a specific antibiotic via intramuscular injection, as prescribed by physicians.

Two intramuscular injections into the right and left Dorsal Gluteal Region (DRG) were recorded for each participant. One was administered by a nurse, according to the unit's routine, and took 5 seconds to complete. A day after, the same nurse gave the other injection in the opposite DGR, taking 40 seconds to administer. The five-second injections were considered the control group, while the 40 seconds injections were the intervention group. The order of interventions was randomized. The pain level was determined and recorded immediately after each injection.

The study was conducted between September 2019 to November 2019 in the emergency unit of an educational hospital in Istanbul. The data was collected using a Demographic Form, Facial Expressions Scale, and Visual Comparison Scale. Statistical analysis was performed using the Kolmogorov-Smirnov test, Mann-Whitney U test, Wilcoxon test, and Spearman correlation analysis, with a significance level of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Having a condition leads to prescribing Clindamycin 600 mg/4 ml intramuscularly Having no pain in the area of injection Absence of any tissue damage history at the site of injection

Exclusion Criteria:

Asking for withdrawal after signing the informed consent Intensifying the disease/condition at the time of the second injection Taking any analgesic medication before the application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Facial Pain Expressions Scale | after implamention in 1-2 seconds
  Between one to ten
Visual Pain Comparison Scale | after implamention in 1-2 seconds
  Six level: Between zero to six

CONTACTS AND LOCATIONS:
Locations (1):
- Leman Şenturan, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided